CLINICAL TRIAL: NCT02520505
Title: Determining the Fertility Benefit of Immediate SO+IUI After Operative Laparoscopy in Patients With Advanced Stage Endometriosis
Brief Title: SO+IUI After Operative Laparoscopy in Patients With Advanced Stage Endometriosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15-149
Record Dates: First submitted 2015-07-11; First posted 2015-08-13 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Endometriosis; Infertility
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Clomiphene; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expectant Management: Timed Intercourse (Other): Patients randomized to expectant management will be counseled on timed intercourse and the window in which intercourse should be performed during the randomization phone call. Patients will be encouraged to contact their fertility doctor and the primary investigator if they become pregnant and an estimated date of confinement will be calculated based upon the patient's last menstrual period. Patients will also be notified that they will be contacted at the end of the six month timeframe to inquire as to whether or not they became pregnant.
  Interventions: Behavioral: Timed intercourse
- Supraovulation + IUI (Active Comparator): Women randomized to super ovulation (SO) will be treated according to a standard protocol under the care of their staff physician and fertility nurses. The patient will be treated with 100mg/day of clomiphene citrate starting on day 3 of the menstrual cycle and ending on day 7. Intrauterine insemination will be performed 36 hours after the hCG surge (follicle rupture) by inserting a catheter through the cervix of the patient in dorsal lithotomy position.
  Interventions: Drug: Supraovulation clomiphene citrate; Procedure: Intrauterine Insemination

INTERVENTIONS:
Drug: Supraovulation clomiphene citrate — Treatment with clomiphene citrate during day 3 to 7 of the menstrual cycle.
  Other Names: Clomiphene citrate
  Arms: Supraovulation + IUI
Behavioral: Timed intercourse — Timing intercourse during the fertile window in the menstrual cycle. Patients may also utilize an ovulation predictor kit to determine time of ovulation.
  Other Names: Expectant management
  Arms: Expectant Management: Timed Intercourse
Procedure: Intrauterine Insemination — Intrauterine insemination will be performed ~36 hours after the time the woman ovulates, as determined by an ovulation predictor kit.
  Other Names: IUI
  Arms: Supraovulation + IUI

SUMMARY:
This is a prospective randomized control, crossover trial to determine if supraovulation with clomiphene citrate and intrauterine insemination is more efficacious than expectant management in women with stage III or IV endometriosis who have recently undergone operative laparoscopy.

DETAILED DESCRIPTION:
This is a prospective randomized control, crossover trial that will be performed examining fertility outcomes in patients after ablative and/or excisional operative laparoscopy at the Cleveland Clinic for infertility due to advanced stage (III/IV) endometriosis. Patients will be randomized to either receive immediate (three months) clomiphene citrate at 100mg daily for SO+IUI or expectant management with timed intercourse for three months. After 3 months, patients will cross over to the other treatment arm, receiving either three additional months of SO+IUI or three months of expectant management. Monthly fecundity rates and additional outcomes will be monitored.

The study population will include women 18 to 35 years old with a diagnosis of infertility, defined as actively attempting to achieve pregnancy for >12 months of unprotected intercourse, prior to undergoing operative laparoscopy to treat endometriosis. Using the ASRM classification criteria, all patients included will have a diagnosis of stage III or IV endometriosis from a surgery performed within the Cleveland Clinic Foundation. Patients who present with idiopathic infertility who are found to have advanced stage endometriosis on diagnostic laparoscopy will be included as long as ablation and/or excision was performed on all visible endometriosis and adhesions. All patients must have at least one patent fallopian tube, assessed by hysterosalpingogram, hysteroscopy, or at the time of laparoscopy via chromopertubation. Patients with additional conditions affecting fertility will be included given the factors are classified as mild. This includes uterine leiomyoma(s) with a normal uterine cavity, polycystic ovarian syndrome, and mild male factor infertility (<15 million but >10 million motile sperm per ejaculate before washing). Patients who pursue IVF after expectant management or SO+IUI will be considered as having a negative pregnancy outcome during their participation in the study.

Exclusion criteria include patients with additional causes for infertility such as male factor (<15 million motile sperm per ejaculate), ovulatory dysfunction, polycystic ovarian syndrome, age >35 years, and septate uterus. Patients who have had hormonal therapy in the three months prior to surgery will also be excluded, as this can impact the staging of disease. Patients will also be excluded from the study if they have previously undergone treatments for infertility, such as ovulation induction, IUI and/or IVF.

Potential study participants will be identified by members of the Fertility Center within the Cleveland Clinic Women's Health Institute, as well as by chart review performed by the research coordinator. Women who present to the Cleveland Clinic for evaluation of infertility and are scheduled to undergo surgical intervention will be evaluated for participation in the study. A thorough chart review will be performed to ensure that all inclusion criteria for the study are met. At this time, a copy of the informed consent will be mailed to any patient who meets the study criteria. The primary investigator will call the patient ~1week after the consent document was sent to discuss the study with the patient. For patients with known stage III or IV endometriosis, contact for enrollment into the study will occur after their preoperative visit. Patients with idiopathic infertility who are found to have stage III or IV endometriosis at the time of laparoscopy will be contacted in a similar fashion in the postoperative period. During the phone conversation with the primary investigator, the informed consent process will be described to the patient. Preferentially, patients will schedule a time to meet with the research coordinator to sign the informed consent document at main campus. A one-time parking validation will be provided for these patients. In an effort to accommodate individuals who are unable to travel to main campus to sign the informed consent, the patient will be permitted to sign the document and return it to main campus by mail. The primary investigator will then sign the document and a copy will be mailed back to the patient. The method by which the patient signed the consent, as well as the time line throughout the consent process will be documented in the patient's Epic chart. After informed consent, patients will be randomly assigned to the initial treatment group in the postoperative period. Patients initially assigned to SO+IUI will have a quantitative hCG level drawn after three weeks after IUI. Patients initially assigned to expectant management will be contacted after 3 months to evaluate whether or not spontaneous pregnancy was achieved. As this is a crossover study, patients who do not achieve pregnancy during their initial treatment arm, cross over will occur and patients will undergo 3 months of the remaining treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Using the ASRM classification criteria, all patients included will have a diagnosis of stage III or IV endometriosis from a surgery performed within the Cleveland Clinic Foundation.
* Patients who present with idiopathic infertility who are found to have advanced stage endometriosis on diagnostic laparoscopy will be included as long as ablation and/or excision was performed on all visible endometriosis and adhesions.
* All patients must have at least one patent fallopian tube, assessed by hysterosalpingogram, hysteroscopy, or at the time of laparoscopy via chromopertubation.
* Patients with additional conditions affecting fertility will be included given the factors are classified as mild. This includes uterine leiomyoma(s) with a normal uterine cavity, polycystic ovarian syndrome, and mild male factor infertility (<15 million but >10 million motile sperm per ejaculate before washing).

Exclusion Criteria:

* Exclusion criteria include patients with additional causes for infertility such as male factor (<15 million motile sperm per ejaculate), ovulatory dysfunction, polycystic ovarian syndrome, age >35 years, and septate uterus.
* Patients who have had hormonal therapy in the three months prior to surgery will also be excluded, as this can impact the staging of disease.
* Patients will also be excluded from the study if they have previously undergone treatments for infertility, such as ovulation induction, IUI and/or IVF.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates in SO+IUI versus expectant management | Patients will participate in the study up to 6 months, starting from the first menstrual period after surgery until the completion of the second three month arm of the study.
  The primary objective of this study is to determine whether or not immediate clomiphene citrate SO+IUI is more efficacious for improving pregnancy rates in patients with stage III/IV endometriosis after operative laparoscopy as compared expectant management.

SECONDARY OUTCOMES:
Post-operative fecundity rates in SO+IUI versus expectant management groups | Patients will participate in the study up to 6 months, starting from the first menstrual period after surgery until the completion of the second three month arm of the study.
  A secondary objective is to determine the post-operative fecundity rates in women with stage III/IV endometriosis as compared to the timed intercourse group.
Patient characteristics in SO+IUI versus expectant management groups | Patients will participate in the study up to 6 months, starting from the first menstrual period after surgery until the completion of the second three month arm of the study.
  A secondary objective is to investigate patient characteristics that may affect pregnancy outcomes.
Time to pregnancy in SO+IUI versus expectant management groups | Patients will participate in the study up to 6 months, starting from the first menstrual period after surgery until the completion of the second three month arm of the study.
  A secondary objective is to estimate the time to pregnancy between SO+IUI and expectant management.
Endometriosis fertility index in SO+IUI versus expectant management groups | Patients will participate in the study up to 6 months, starting from the first menstrual period after surgery until the completion of the second three month arm of the study.
  A secondary objective is to determine whether or not the endometriosis fertility index has an impact on outcomes between SO+IUI and expectant management.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Hickman, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States